CLINICAL TRIAL: NCT01982799
Title: Local Anesthesia and Analgesics in Post-Operative Endodontic Pain
Brief Title: Local Anesthesia and Analgesics in Endodontic Pain
Acronym: LAAEP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough funding
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22245
Record Dates: First submitted 2013-10-31; First posted 2013-11-13 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Odontalgia
Keywords: Endodontic treatment, analgesics, anesthesia, post-operative pain
MeSH Terms: conditions — Toothache; Pain, Postoperative | interventions — Ibuprofen; Naproxen; Acetaminophen; Hydrocodone; acetaminophen, hydrocodone drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endododontic Tx + Long acting local anesthetic (Experimental): long acting local anesthetic
  Interventions: Drug: Oral placebo; Drug: Oral ibuprofen; Drug: oral naproxen; Drug: oral acetaminophen/hydrocodone + ibuprofen
- Endodontic Tx plus local anesthetic (Experimental): local anesthetic
  Interventions: Drug: Oral placebo; Drug: Oral ibuprofen; Drug: oral naproxen; Drug: oral acetaminophen/hydrocodone + ibuprofen

INTERVENTIONS:
Drug: Oral placebo — placebo
Drug: Oral ibuprofen — Ibuprofen
Drug: oral naproxen — naproxen
Drug: oral acetaminophen/hydrocodone + ibuprofen — vicodin/ibuprofen
  Other Names: Vicodin plus ibuprofen

SUMMARY:
For patients with a toothache, is pain relief after root canal procedure improved using long acting local anesthetic and analgesics? The purpose of this clinical trial is the investigate the effect of long acting local anesthetic with 1 of 4 oral medication groups, on post-operative endodontic pain.

DETAILED DESCRIPTION:
Patients (n=220) presenting to the University of Minnesota Endodontic clinic, with moderate to severe pain from toothache requiring root canal treatment ,will be invited to participate in the study. The endodontic treatment is NOT part of the research. Patients will complete pain evaluation forms and take 2 doses of prescribed medication. Normally after a root canal procedure, patients will be suggested to take over-the-counter ibuprofen if needed, or prescribed an analgesic if they are having severe pain. We will be randomizing patients in double blind manner to receive regular or long acting local anesthesia and post-op medications (placebo or 1 of 3 analgesics), with the patient evaluating their pain before starting root canal (pre-treatment pain), after root canal, after analgesics and during the following day.

ELIGIBILITY:
Inclusion Criteria:

18-65 y.o. American Society of Anesthesiologists physical classification I or II Can understand and complete pain evaluation forms tooth pain (>3 out of 10) needing root canal Ability to read and provide informed consent Must be able to swallow tablets

Exclusion Criteria:

Allergy/intolerance to analgesics (ibuprofen, naproxen, vicodin) Patients who are pregnant Patients currently on pain medications for an unrelated condition Patients unwilling to fill out pain scales Liver or kidney disease Unable to understand and complete consent form and pain evaluation forms

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Effect of long acting anesthesia and analgesics on endodontic pain | 36 hours
  Pain evaluation time points - pretreatment, after endodontic treatment, 2 hrs after analgesic dosing, following day

SECONDARY OUTCOMES:
Effect of gender and age on post-operative endodontic pain treatment | 36 hours
  Effect of gender and age will be evaluated based on data from pain evaluation forms

CONTACTS AND LOCATIONS:
Overall Officials: Walter Bowles, DDS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota School of Dentistry, Minneapolis, Minnesota, United States